CLINICAL TRIAL: NCT00124163
Title: CT Colonography Ph. I CDI Trial: Evaluation of Stool Tagging for Improved Patient Compliance
Brief Title: Evaluation of Stool Tagging for Improved Patient Compliance
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Center for Diagnostic Imaging (Other)
Other Study IDs: 633
Record Dates: First submitted 2005-07-25; First posted 2005-07-27 (Estimated); Last update posted 2006-02-02 (Estimated); Status verified 2006-01

CONDITIONS: Colon Cancer; Polyps
Keywords: CT Virtual Colonoscopy; Optical Colonoscopy; Stool Tagging; Patient Preparation
MeSH Terms: conditions — Colonic Neoplasms; Polyps

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Procedure: Imaging procedure of CT colonography

SUMMARY:
Computed tomography (CT) colonography has gained widespread multi-disciplinary interest as an evolving noninvasive colorectal screening examination, with the potential of improved patient compliance. The investigator's prior work demonstrated that the bowel preparation was the least tolerable aspect of colorectal evaluation when compared to the CT colonography and optical colonoscopy procedures. Stool tagging could provide a more gentle and efficient bowel preparation, with fewer false positives due to retained stool-mimicking polyps.

The researchers hypothesize that image quality and patient preference will vary with stool tagging concentration and dosing schedule. The researchers propose to evaluate specific stool tagging protocols with the following aims:

AIM 1: Perform a randomized trial of three specific stool tagging protocols using barium and iodine at CT colonography in a well-characterized cohort of patients undergoing colorectal evaluation.

AIM 2: Analyze the CT colonography and optical colonoscopy data to assess differences across stool tagging protocols for the outcome measures of patient preference, image quality in the presence of tagging, and diagnostic reader performance.

The researchers will use specific variations in stool tagging techniques to determine the best image quality of CT data (e.g., homogenous tagging of fluid and stool), and highest patient acceptability, as well as evaluate the adequacy of preparation for same-day colonoscopy. Diagnostic reader performance will focus on the accuracy for detecting all neoplastic lesions including colon cancers, adenomatous polyps, sessile adenomas and flat adenomas. Most importantly, these results will help inform the design of a larger trial of an optimized CT colonography technique in a community setting.

DETAILED DESCRIPTION:
CT Colonography, a rapidly evolving technique, offers a noninvasive and efficient colorectal screening examination, with the potential to improve patient compliance. However, currently it requires the bowel preparation, one of the largest barriers to colonoscopy screening. A promising new tool in CT Colonography is stool tagging, which has the potential to decrease the amount of catharsis required by patients during the bowel preparation, while decreasing the number of false positives due to the reader mistaking residual stool for polyps.

Our primary hypothesis is that image quality and patient compliance differ depending upon the tagging agent and dosing schedule. Our strategy is to vary key components of recently reported barium and iodine protocols to further optimize them and to compare our results with existing and currently aggregating data in collaboration with other investigators.

The following aims will implement this strategy:

AIM 1: Perform a randomized control trial of specific stool tagging protocols at CT Colonography in a well characterized cohort of patients undergoing colorectal evaluation.

Task 1A - Recruit a prospective cohort of 60 subjects, randomize them equally to three different stool tagging protocols, and sequentially perform CT Colonography and optical colonoscopy on them.

Task 1B - Assess image quality of CT Colonography and optical colonoscopy data by the method of bowel preparation in the first five subjects of each arm and implement specific changes, if necessary.

AIM 2: Analyze the CT Colonography and optical colonoscopy data to assess differences across study arms for the outcome measures of patient preference, image quality of tagged stool, and diagnostic reader performance.

Task 2A: Assess patient expectations regarding the bowel preparations, CT Colonography and colonoscopy before the procedures and their preferences after the procedures.

Task 2B: Evaluate image quality, in the presence of tagged stool and fluid, of both the CT data and the colonoscopy data.

Task 2C: Perform a multi-observer reader evaluation of diagnostic performance of CT Colonography and colonoscopy, compared to the enhanced reference standard of colonoscopy aided by segmental unblinding of CT results, to assess sensitivity and specificity of colorectal polyp detection.

Upon completion, the three specific variations in stool tagging techniques will be compared on homogenous density of tagging and patient acceptability to determine which protocol optimizes the trade-off. Diagnostic performance of CT and colonoscopy will be compared to the enhanced reference standard of colonoscopy aided by the segmental unblinding of CT results. Most significantly, these results may help determine an optimal tagging protocol to use for larger trials of CT Colonography implementation in community settings.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are 45 to 80 years old for routine screening colonoscopy

Exclusion Criteria:

* Patients with inflammatory bowel disease
* Patients with polyposis syndromes
* Pregnant women
* Patients over 350 pounds
* Patients with bright red blood per rectum
* Patients who have a contraindication to undergo outpatient colonoscopy, including patients on blood thinners, prior myocardial infarction (MI) in the last six months, history of congestive heart failure (CHF), history of arrhythmia, patients too weak to transfer themselves from a bed to a chair, or patients with severe constipation who would require a two day bowel preparation.

All subjects will undergo informed consent by the St. Luke's institutional review board (IRB). Referred subjects will be asked if they are interested in the study and those responding affirmatively will be transferred to a recruiter to learn about the study and begin the consent process if interested.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2005-07

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth G. McFarland, MD, Principal Investigator — St. Luke's Hospital
Locations (1):
- Diagnostic Imaging Associates, Chesterfield, Missouri, United States

REFERENCES:
- [Background] Pickhardt PJ, Choi JR, Hwang I, Butler JA, Puckett ML, Hildebrandt HA, Wong RK, Nugent PA, Mysliwiec PA, Schindler WR. Computed tomographic virtual colonoscopy to screen for colorectal neoplasia in asymptomatic adults. N Engl J Med. 2003 Dec 4;349(23):2191-200. doi: 10.1056/NEJMoa031618. Epub 2003 Dec 1. PMID 14657426
- [Background] Iannaccone R, Laghi A, Catalano C, Mangiapane F, Lamazza A, Schillaci A, Sinibaldi G, Murakami T, Sammartino P, Hori M, Piacentini F, Nofroni I, Stipa V, Passariello R. Computed tomographic colonography without cathartic preparation for the detection of colorectal polyps. Gastroenterology. 2004 Nov;127(5):1300-11. doi: 10.1053/j.gastro.2004.08.025. PMID 15520999
- [Background] Lefere PA, Gryspeerdt SS, Dewyspelaere J, Baekelandt M, Van Holsbeeck BG. Dietary fecal tagging as a cleansing method before CT colonography: initial results polyp detection and patient acceptance. Radiology. 2002 Aug;224(2):393-403. doi: 10.1148/radiol.2241011222. PMID 12147834